CLINICAL TRIAL: NCT06581250
Title: No-Show Prevention Practices in Dental Care Settings Serving Underserved Populations
Brief Title: Improving Show Rates in Dental Care Settings Serving Underserved Populations
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 2024-1502; 4UH3DE030531-03 (NIH); A195010 (Other: UW Madison); 2024-1086 (Other: Previous IRB number)
Record Dates: First submitted 2024-08-22; First posted 2024-09-03 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Dental Care
Keywords: Patients That Don't Attend Appointments; Dental Patients; No-Show; Underserved

STUDY DESIGN:
Intervention Model Description: The study uses a 2x2x2 factorial cluster-randomized design The unit of intervention and randomization will be dental clinic sites (clusters). Forty clinics will be randomized between eight possible combinations of receiving or not receiving the three study interventions. The factorial structure of the design ensures that 20 clinic sites receive each intervention, and 20 do not. Five clinic sites will receive none of the interventions, five clinics will receive all three interventions, and 30 clinic sites will receive a different combination of 2 of the 3 interventions.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Control (No Intervention)
- Reminder Messages (Active Comparator)
  Interventions: Behavioral: Reminder Messages
- Walk-in Visits (Active Comparator)
  Interventions: Behavioral: Walk-in Visits
- Motivation-enhanced Communication (Active Comparator)
  Interventions: Behavioral: Motivation-enhanced Communication
- Reminder Messages & Walk-in visits (Active Comparator)
  Interventions: Behavioral: Reminder Messages; Behavioral: Walk-in Visits
- Reminder Messages & Motivation-enhanced Communication (Active Comparator)
  Interventions: Behavioral: Reminder Messages; Behavioral: Motivation-enhanced Communication
- Walk-in visits & Motivation-enhanced Communication (Active Comparator)
  Interventions: Behavioral: Walk-in Visits; Behavioral: Motivation-enhanced Communication
- Reminder Messages, Walk-in visits, & Motivation-enhanced Communication (Active Comparator)
  Interventions: Behavioral: Reminder Messages; Behavioral: Walk-in Visits; Behavioral: Motivation-enhanced Communication

INTERVENTIONS:
Behavioral: Reminder Messages — Dental clinic staff will use scripts to contact patients 24 and 48 hours before appointments. These scripts will guide staff in confirming the patient will appear for their appointment.
  Arms: Reminder Messages; Reminder Messages & Motivation-enhanced Communication; Reminder Messages & Walk-in visits; Reminder Messages, Walk-in visits, & Motivation-enhanced Communication
Behavioral: Walk-in Visits — When contacting patients to schedule an appointment (by phone, email, text, or other methods), dental clinic staff will notify patients of times during which patients can walk-in for a dental visit, if convenient for them; otherwise, a regular appointment will be arranged. Scheduled appointments will continue to be available in addition to the walk-in hours.
  Arms: Reminder Messages & Walk-in visits; Reminder Messages, Walk-in visits, & Motivation-enhanced Communication; Walk-in Visits; Walk-in visits & Motivation-enhanced Communication
Behavioral: Motivation-enhanced Communication — Participating clinic site staff will be trained in motivation-enhanced communication techniques using the guide for dental clinic sites and coaching. Topics to be included in the motivation-enhanced communication training are a) to determine what patients hope to gain from their dental care, steps needed to succeed, how the agency and client will work together to attain the goals, and b) to identify patient barriers to attending their visit (e.g., transportation, payment, do not understand need for visit, etc.), and what the agency and patient will do to overcome those barriers. Staff will be instructed to use these techniques with patients at every contact about an upcoming appointment.
  Arms: Motivation-enhanced Communication; Reminder Messages & Motivation-enhanced Communication; Reminder Messages, Walk-in visits, & Motivation-enhanced Communication; Walk-in visits & Motivation-enhanced Communication

SUMMARY:
The goal of this study is to compare different no-show interventions in dental clinics serving underserved populations. The main question it seeks to answer is

* How do different no-show intervention methods compare in reducing no-shows?

Participants will be asked to

* Implement different interventions
* Report a limited set of data to researchers

DETAILED DESCRIPTION:
Persistent no-show rates contribute to the oral health disparities and inadequate access to dental care that disproportionately affect underserved populations. The proposed research will test the impact of three different strategies on improving show rates using a full factorial design. Specifically, the study is designed as a 2×2×2 factorial cluster-randomized trial of reminder messaging, motivation-enhanced communication, and walk-in visit. The unit of intervention and randomization will be dental clinic sites (clusters). Forty clinics will be randomized between eight possible combinations of receiving or not receiving the three study interventions, with five clinics receiving each intervention. Findings from this study seek to provide an evidence-based approach to reducing no-shows and increasing access to dental care for underserved populations.

ELIGIBILITY:
Inclusion Criteria:

Sites must be:

* Serve at least a 51 percent self-pay and Medicaid patients
* Be willing to provide limited data sets of clinic data to the research team
* Be willing to undertake and support and organizational improvement project to improve show rates

Staff must be:

* A paid staff member at a participating clinic
* Be able and willing to provide written or verbal consent

Exclusion Criteria:

* No exclusion criteria for clinics or staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-04 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in proportion of scheduled appointments for which the patient attends, pre-to-post intervention | 6 months pre-intervention to 12 months post-intervention
  To test the efficacy of motivation-enhanced communication, reminder messaging, and walk-in visits as compared to treatment as usual For each of the three interventions, the pre-to-post intervention change in show rates.
  Show rate is defined as the proportion of scheduled appointments for which the patient attends their scheduled clinic appointment. Appointments cancelled or rescheduled more than 24 hours in advance are not included in the calculation.
  Outcome will be measured by data exported from the clinical electronic health records monthly.

SECONDARY OUTCOMES:
Organizational Change Manager (OCM) Score | Survey will be administered at 3 months
  To examine whether Organizational Readiness for Change moderates the efficacy of the targeted evidence-based practices.
  Organizational readiness for change will be assessed by a validated 16-item index called the Organizational Change Manager (OCM) For each clinic site, a group of 5 people that includes clinicians, dental hygienists, manager, and scheduler each team member will provide their own OCM responses.
  Outcome will be measured by combined responses to Organizational Change Manager survey tool. Total possible ranges of scores will be 0-104, with a higher score indicating increased readiness. The responses to the Organizational Change Manager survey from each clinic staff respondent will be added and an average of those scores will be calculated.
Statistical Comparison of Interventions for Effectiveness Analysis | 6 months pre-intervention to 12 months post-intervention
  Evaluate the efficacy of motivation-enhanced communication, reminder messaging, and walk-in visits compared to each other.
  Comparative effectiveness analyses: Evaluate the efficacy of motivation-enhanced communication, reminder messaging, and walk-in visits compared to each other For each of the interventions, the difference in the pre-to-post intervention change in show rates in clinics receiving the different interventions Outcomes will be measured by data exported from the clinical electronic health records monthly.
Statistical Comparison of Combining Multiple Interventions for Interaction Analysis | 6 months pre-intervention to 12 months post-intervention
  Evaluate the synergy of combining multiple interventions. For each pair of interventions, the difference in the pre-to-post intervention change in show rates in clinics receiving both interventions compared to clinics receiving only one of them.
  Outcomes will be measured by data exported from the clinical electronic health records monthly.

CONTACTS AND LOCATIONS:
Overall Officials: Todd Molfenter, PhD, Principal Investigator — University of Wisconsin, Madison; Chris Okunseri, BDS, MSc, MLS, DDPHRCSE, Principal Investigator — Marquette University
Locations (1):
- University of Wisconsin - Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No